CLINICAL TRIAL: NCT03774212
Title: Do Active Noise Cancelling Headphones With White Noise Masking Improve Sleep in Non-ventilated, Non-delirious Critical Care Patients?
Brief Title: Sleep Headphones and HDU: a Novel Intervention and Sound Evaluation
Acronym: SHH: Noise!
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AC18134
Record Dates: First submitted 2018-12-07; First posted 2018-12-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Sleep Deprivation; Sleep
Keywords: Critical care patients; High dependency unit; Intensive care unit
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): On study night 1, participants will receive standard care (no headphones provided). On study night 2, these patients will wear Active Noise Cancelling headphones playing white noise.
  Interventions: Device: Active noise cancelling headphones
- Group B (Experimental): Patients will spend night 1 wearing Active Noise Cancelling headphones playing white noise. On Study night 2, these patients will receive standard care (no headphones provided).
  Interventions: Device: Active noise cancelling headphones

INTERVENTIONS:
Device: Active noise cancelling headphones — The white noise will play from an 'iPod touch' (Apple), through the active noise cancelling headphones.
  Other Names: White noise masking

SUMMARY:
It is well established that patients sleep poorly in the Intensive Care Unit (ICU), and excessive noise is considered to be a modifiable cause of this. Previous studies have tried to reduce ambient noise by educating staff and fixing noisy equipment. Other studies have tried to reduce the noise experienced by patients by supplying them with active noise cancelling headphones and earplugs. In this study we are combining Active Noise Cancelling headphones with white noise to try and reduce noise experienced by patients, with the aim of improving their sleep. Sleep deprivation is known to negatively impact health, and so improving sleep may improve patient outcomes as well as improve the patient's experience in critical care.

The Investigators will screen all patients in the critical care wards in the Royal Infirmary of Edinburgh. Patients that are receiving ventilation, are delirious or have already been enrolled in the study will be excluded. After allowing patients to give informed consent, we will randomise them into one of two study groups:

Study group A will receive standard care on the 1st night (no headphones), and will receive the intervention (active noise cancelling headphones with white noise) on the 2nd night.

Study group B will receive the intervention on the 1st night, and will receive standard care on the 2nd night.

All patients will wear a Xiaomi MiBand 2 wrist band, that tracks movement and sleep.

Patients will fill in the Pittsburgh Sleep Quality Index at the beginning of the study to establish usual sleeping habits.

Our primary outcome measure is the mean score on the Richard Campbell Sleep Questionnaire (RCSQ), which will be filled in by the patient the morning after each night.

Our secondary outcome measure is the data from the wrist band, noise levels measured overnight, and patient experience of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Critical care patient in Royal Infirmary of Edinburgh

Exclusion Criteria:

* < 18 years of age
* If the patient is delirious. This will be clarified by asking the nurses, who use the Confusion Assessment method for the ICU (CAM-ICU) Score.
* If the patient is receiving any form of ventilation (invasive or non-invasive ventilation, continuous positive airway pressure (CPAP), High flow nasal oxygen (HFNO) or respiratory support at night)
* Physical reasons why they can't wear over-ear headphones
* Pre-existing severe hearing impairment
* Previous participation in the study.
* If the patient is likely to receive medical interventions during the night that would disturb their sleep.
* Patients expected to leave the critical care wards within the following 48hours.
* Refusing consent or inability to give consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-03-18 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in score on the Richards-Campbell sleep questionnaire. | Day 1 and day 2 after participant's enrolment. Completed throughout the 6 month study duration.
  Richards-Campbell sleep questionnaire is a series of 5 Visual analog scales that are 100mm long, and range from "best possible" to "worst possible". The final result is calculated by taking a mean of the distances along each line (from left to right).

SECONDARY OUTCOMES:
Patient experience | Day 2 after participant's enrolment. Completed throughout the 6 month study duration.
  Patients will fill out a questionnaire about their experience. Participants will be required to circle an appropriate descriptive word to answer each question.
Actigraphy data | Night 1 and 2 of participant's enrolment. Completed throughout the 6 month study duration.
  The wrist band provides:
  * Total sleep time
  * Deep sleep time
  * Light sleep Time

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data with other researchers